CLINICAL TRIAL: NCT05456997
Title: Prospective Observational Study of Metabolic Myopathy in Cushing's Syndrome or Pheochromocytoma Patients Undergoing Adrenalectomy
Brief Title: Metabolic Myopathy in Endocrinopathy
Acronym: LYDIA
Status: Terminated | Type: Observational
Why Stopped: Loss of research capable staff
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Imperial College London (Other); Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: Pending
Record Dates: First submitted 2022-05-04; First posted 2022-07-13 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2022-04

CONDITIONS: Cushing Syndrome; Pheochromocytoma; Conns Syndrome; Metabolic Myopathy
Keywords: Epigenetic control
MeSH Terms: conditions — Cushing Syndrome; Pheochromocytoma; Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Abdominal wall muscle biopsy Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cushings syndrome: Patients with Cushing's syndrome treated medically prior to adrenalectomy
  Interventions: Procedure: Muscle biopsy
- Phaeochromocytoma and paraganglioma (PPGL): Patients with PPGL treated medically prior to adrenalectomy
  Interventions: Procedure: Muscle biopsy
- Conn's syndrome: Patients with Conn's syndrome treated medically prior to adrenalectomy
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — Patients will have muscle biopsies taken at time of surgery under general anaesthetic. Open biopsies from the operation field (abdominal wall) will be taken by the surgical team without extending or making new skin incisions. Briefly, muscle samples (approximately 0.5cm3) are excised and haemostasis secured. The muscle biopsies will be snap frozen and stored at -80°C for the analysis of pathways relevant to muscle homeostasis using biochemical and molecular techniques.

SUMMARY:
Endocrine diseases including Cushing's syndrome and phaeochromocytoma/paraganglioma (PPGL) but not Conn's syndrome are associated with muscle wasting and weakness. The study's aim is to identify epigenetic determinants of muscle homeostasis in these conditions following medical treatment and adrenalectomy. This is an observational pilot study that will recruit 66 patients from 3 diagnostic groups: Cushing's syndrome (16), PPGL (20) and Conn's syndrome (30). Indices of muscle bulk and strength will be assessed at diagnosis and at outpatient follow-up 6-9 weeks after adrenalectomy. At these times blood and urine will be collected and a muscle biopsy taken from the operation site at the time of surgery. Pathway analysis in these samples will identify potentially novel signalling pathways contributing to muscle wasting via prolonged exposure to high levels of corticosteroid and catecholamines. This will highlight commonalities and differences in pathogenesis of muscle wasting from a variety of different causes. Finally, it will inform identification of novel therapies for muscle atrophy.

DETAILED DESCRIPTION:
Muscle wasting and weakness is important because it accounts for a large proportion of the disability associated with disease and normal aging. The annual economic cost in the USA alone has been estimated at $1.8 billion.

The investigators have studied muscle wasting associated with chronic and acute illness, finding a marked dissociation between wasting and disease severity. This indicated that epigenetic and genetic factors may contribute to individual susceptibility to wasting. To analyse factors controlling muscle mass, the investigators have developed a novel clinical model of muscle loss. Hence, in patients undergoing aortic surgery, a large insult is imposed on patients with a background of a disease that leads to muscle wasting (reduced cardiac function). As the timing of the insult is known, the investigators can follow muscle wasting longitudinally. Our recent work using this model has characterised novel muscle signalling pathways that mediate muscle breakdown. Specifically, the investigators found that 50% of patients undergoing cardiac surgery lose significant muscle mass (>10% in the "wasters" group) in the 7 days after uncomplicated surgery, which correlated with loss of strength 7-9 Expression of microRNAs (miRNAs) from imprinted loci (C19MC miRNAs and miR-675) in muscle biopsy samples was strongly associated with subsequent muscle wasting and weakness. Furthermore, expression of these miRNA in myoblasts and animal models confirms their effects on muscle and suggests modes of action through transforming growth factor signalling pathways, ribosome assembly and mitochondrial function. Finally, metabolomic analysis of plasma samples from these patients suggested that exposure to higher levels of active intrinsic corticosteroid, a known cause of sarcopenia, was correlated with muscle loss. Acute muscle wasting (ICU acquired weakness) is associated with high levels of corticosteroids, owing to a defect in deactivation, and shock which is countered with high doses of catecholamines. The investigators will measure miR expression, and longitudinal muscle bulk and strength in patients undergoing adrenalectomy at SBH.

Group 1: Cushing's syndrome caused by very elevated levels of corticosteroids, associated with severe wasting.

Group 2: Phaeochromocytoma and paraganglioma (PPGL) caused by very elevated levels of catecholamines, associated with moderate wasting.

Group 3: Conn's syndrome caused by elevated mineralocorticoid, not associated with muscle wasting (Control group) All patients will be assessed at diagnosis, after medical treatment and after completed reversal of the defect after surgery. Various measures of focal and global strength and function will be recorded alongside measures of muscle bulk. A muscle biopsy from the wound site will be taken at surgery.

One of the key epigenetic determinants of muscle wasting in acute and chronic conditions is micro-RNA (miR-) 424, which targets ribosome synthesis and function as well as insulin sensitivity. The promotor for its' large non-coding RNA precursor contains a steroid responsive region. Therefore overall, the investigators expect miR-424 expression to be correlated with muscle wasting across the 3 patient groups. Mi-RNA profiles will be generated in patient blood and muscle samples: our previous studies have shown that muscle expression of selected mi-RNA is a strong predictor of the response to injury and in patients with chronic respiratory failure (COPD) corresponding circulating levels can be measured in contemporaneous blood samples.

A predictive biomarker (miR expression in blood) would allow a personalised approach to clinical trials for anti-muscle atrophy therapies. The miRNA profiles in blood associated with muscle wasting are likely to be useful predictive biomarkers for several conditions associated with sarcopenia, as evidenced by previous miRNA sets associating with muscle phenotype in COPD and in patients undergoing cardiac surgery.

Pathway analysis will identify potentially novel signalling pathways contributing to muscle wasting via prolonged exposure to high levels of corticosteroid or increased inflammatory sensitivity. This will highlight commonalities and differences in pathogenesis of muscle wasting from a variety of different causes. Finally, it will inform identification of novel therapies for muscle atrophy.

Insensitivity to insulin is a hallmark of many acute and chronic diseases, and a feature of metabolic syndrome. The investigators will be able to determine the potential role of high circulating levels of miR-424, which could constitute a novel therapeutic approach to type 2 diabetes. Similarly, owing to the multi-system insult of cardiac surgery our patient cohorts suffered acute kidney injury and systemic inflammation requiring vasopressors. These data have been collected and could be mined in the future to identify epigenetic determinants and pathways associated with these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* Receiving both medical management and adrenalectomy for treatment of Cushing's syndrome or phaeochromocytoma at St Bartholomew's Hospital (SBH)

Exclusion Criteria:

* Previous Stroke
* Neuromuscular disease
* Disseminated Malignancy
* Underlying neuromuscular disease
* Paediatrics
* Non-consenting adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria include any consenting adult receiving adrenalectomy surgery for Cushing's or Conn's syndrome or phaeochromocytoma/ paraganglioma (PPGL) at St Bartholomew's Hospital with no evidence of pre-hospital neuromuscular conditions.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in cross sectional area of the Rectus Femoris (RFcsa) | Day 0/ at presentation to 6-9 week follow up.
  RFcsa will be calculated using B-mode ultrasound (US) at pre-determined time points
Change in Hand Held Dynamometry strength (grip strength) | Day 0/ at presentation to 6-9 week follow up.
  Hand-held dynamometry will be assessed in both hands (the maximum of 3 attempts)
Change in Knee straightening dynamometry | Day 0/ at presentation to 6-9 week follow up.
  The test will be conducted using a Lafayette Manual Muscle Tester. Joint knee moment (torque) and strength will be measured.
Change in Short Physical Performance Battery (SPPB) | Day 0/ at presentation to 6-9 week follow up.
  SPPB is a measure of patients' functional status: scores range from 0 (worst performance) to 12 (best performance).
Change in Lying and Standing Vital Capacity (FVC - forced vital capacity) ratio | Day 0/ at presentation to 6-9 week follow up.
  Lying and standing vital capacity will be measured using a hand held spirometer
Change in bio-impedance indices of body composition | Day 0/ at presentation to 6-9 week follow up.
  Indices of body composition will be measured by electrical impedance.
Change in rectus femoris pixel intensity | Day 0/ at presentation to 6-9 week follow up.
  Pixel intensity is a measure of muscle quality measured by B mode ultrasound

SECONDARY OUTCOMES:
Changes in plasma markers of muscle homeostasis by enzyme-linked immunosorbent assay (ELISA) | Day 0/ at presentation & 6-9 week follow up.
  Insulin-like growth factor-1
Changes in plasma markers of muscle homeostasis by enzyme-linked immunosorbent assay (ELISA) | Day 0/ at presentation & 6-9 week follow up.
  growth and differentiation factor-15
Changes in plasma markers of muscle homeostasis by enzyme-linked immunosorbent assay (ELISA) | Day 0/ at presentation & 6-9 week follow up.
  resistin
Changes in steroid metabolism by mass spectroscopy in blood and urine | Day 0/ at presentation to 6-9 week follow up.
  cortisol: cortisone ratio
Assay in abdominal muscle of markers of muscle atrophy by western blot | Intra-operatively during adrenalectomy
  Atrogen
Assay in abdominal muscle of markers of muscle atrophy by western blot | Intra-operatively during adrenalectomy
  MURF
Unbiased RNA sequencing and targetted qPCR for micro RNAs | Intra-operatively during adrenalectomy
  Assays undertaken on abdominal muscle
Changes in circulating micro-RNAs | Day 0/ at presentation to 6-9 week follow up.
  Unbiased RNA sequencing of plasma samples and targetted qPCR for micro RNAs
Changes in biomarkers of myolysis in urine | Day 0/ at presentation to 6-9 week follow up.
  Assays for histidine
Changes in the metabolome | Day 0/ at presentation to 6-9 week follow up.
  Mass spectroscopy based unbiased metabolic screen in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Griffiths, MB BS, Principal Investigator — Bartshealth NHS Trust
Locations (1):
- Barts Heart Centre, London, County (optional), United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloch SA, Donaldson AV, Lewis A, Banya WA, Polkey MI, Griffiths MJ, Kemp PR. MiR-181a: a potential biomarker of acute muscle wasting following elective high-risk cardiothoracic surgery. Crit Care. 2015 Apr 7;19(1):147. doi: 10.1186/s13054-015-0853-5. PMID 25888214
- [Background] Kemp PR, Griffiths M, Polkey MI. Muscle wasting in the presence of disease, why is it so variable? Biol Rev Camb Philos Soc. 2019 Jun;94(3):1038-1055. doi: 10.1111/brv.12489. Epub 2018 Dec 26. PMID 30588725
- [Background] Donaldson A, Natanek SA, Lewis A, Man WD, Hopkinson NS, Polkey MI, Kemp PR. Increased skeletal muscle-specific microRNA in the blood of patients with COPD. Thorax. 2013 Dec;68(12):1140-9. doi: 10.1136/thoraxjnl-2012-203129. Epub 2013 Jun 28. PMID 23814167
- [Background] Connolly M, Paul R, Farre-Garros R, Natanek SA, Bloch S, Lee J, Lorenzo JP, Patel H, Cooper C, Sayer AA, Wort SJ, Griffiths M, Polkey MI, Kemp PR. miR-424-5p reduces ribosomal RNA and protein synthesis in muscle wasting. J Cachexia Sarcopenia Muscle. 2018 Apr;9(2):400-416. doi: 10.1002/jcsm.12266. Epub 2017 Dec 7. PMID 29215200
- [Background] Kemp PR, Paul R, Hinken AC, Neil D, Russell A, Griffiths MJ. Metabolic profiling shows pre-existing mitochondrial dysfunction contributes to muscle loss in a model of ICU-acquired weakness. J Cachexia Sarcopenia Muscle. 2020 Oct;11(5):1321-1335. doi: 10.1002/jcsm.12597. Epub 2020 Jul 16. PMID 32677363
- [Background] Garros RF, Paul R, Connolly M, Lewis A, Garfield BE, Natanek SA, Bloch S, Mouly V, Griffiths MJ, Polkey MI, Kemp PR. MicroRNA-542 Promotes Mitochondrial Dysfunction and SMAD Activity and Is Elevated in Intensive Care Unit-acquired Weakness. Am J Respir Crit Care Med. 2017 Dec 1;196(11):1422-1433. doi: 10.1164/rccm.201701-0101OC. PMID 28809518
- [Background] Ferrau F, Korbonits M. Metabolic comorbidities in Cushing's syndrome. Eur J Endocrinol. 2015 Oct;173(4):M133-57. doi: 10.1530/EJE-15-0354. Epub 2015 Jun 9. PMID 26060052